CLINICAL TRIAL: NCT05606978
Title: The Effectiveness of Blended Forensic Ambulant Systemic Therapy (FASTb): A Randomized Controlled Trial Comparing Blended and Regular FAST
Brief Title: The Effectiveness of Blended Forensic Ambulant Systemic Therapy
Acronym: FASTb
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Utrecht University (Other)
Collaborators: De Waag (Unknown)
Responsible Party: Principal Investigator, Marjolein van Cappellen, PhD candidate, Utrecht University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 60-63600-98-1138
Record Dates: First submitted 2022-10-25; First posted 2022-11-07 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Conduct Disorder; Antisocial Behavior; Behavioral Disorder
MeSH Terms: conditions — Conduct Disorder; Antisocial Personality Disorder; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FASTb (Experimental): Participants receive FAST blended (FASTb): a combination of face-to-face and online therapy
  Interventions: Behavioral: FASTb
- FASTr (Active Comparator): Participants receive FAST regular (FASTr): face-to-face therapy
  Interventions: Behavioral: FASTr

INTERVENTIONS:
Behavioral: FASTb — FAST blended
  Arms: FASTb
Behavioral: FASTr — FAST regular
  Arms: FASTr

SUMMARY:
The purpose of this study is to investigate whether blended Forensic Ambulant Systemic Therapy (FASTb) is equally effective as regular FAST (FASTr).

DETAILED DESCRIPTION:
Forensic Ambulant Systemic Therapy (FAST) is a promising treatment for juveniles aged 12-21 showing antisocial behavior and conduct disorders. Next to regular FAST (FASTr), a blended version was developed (FASTb), in which face-to-face contact is replaced by minimally 50% online contact over the duration of intervention, consisting of video-calls and eHealth modules. The primary aim of the current study is to investigate whether FASTb is equally effective as FASTr. All clients (and their caregivers) who meet the inclusion and eligibility criteria and who signed informed consent will be assigned to either the FASTr or FASTb condition. Randomization will be done on the family level and will not depend on therapist or treatment site.

ELIGIBILITY:
Every juvenile and caregiver who meets the FAST inclusion criteria is considered for the study. FAST therapists determine whether clients meet the inclusion criteria during the standard FAST intake procedure. The inclusion criteria are:

1. Juvenile has an estimated IQ-score of 80 or higher and/or sufficient adaptive skills to benefit from the intervention. The estimated IQ-score is measured using the Screener voor intelligentie en licht verstandelijke beperking (SCIL). The score on the SCIL determiners whether an IQ-test and/or a measurement of adaptive skills using the ADAPT is necessary;
2. Juvenile is aged 12-21 years old at intervention start;
3. Juvenile exhibits externalizing behavior that results in problems in at least two areas of life (family, school, leisure time), determined by referrer information and/or intake;
4. Juvenile has a medium to high recidivism risk, measured by the Risicotaxatie-instrument voor de Ambulante Forensische GGZ Jeugd (RAF GGZ Jeugd) and/or the Landelijk Instrumentarium Jeugdstrafrechtketen (LIJ);
5. Presence of juvenile-caregiver relationship problems, as measured by the RAF GGZ Jeugd;
6. Juvenile has a diagnosis of a DSM-5 behavioral disorder, which is determined using case file analysis or a new diagnostic process;
7. Caregiver(s) and juvenile cannot be motivated to follow treatment at the outpatient clinic;
8. Juvenile and caregiver(s) have sufficient Dutch language skills, as estimated by the FAST therapist team;
9. Treatment can be offered in either a voluntary or mandatory framework;
10. Juvenile resides with their caregiver(s) or is expected to return to residing with caregiver(s) within the first two months of intervention.

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Clients meet the FAST exclusion criteria, which are:

   1. Juvenile exhibits severe psychiatric symptoms requiring admission;
   2. Problem behavior of the juvenile is caused by primary substance abuse problems;
   3. Caregiver(s) refuse structurally to participate in treatment
   4. The safety of the therapist or family members cannot be guaranteed sufficiently;
2. Clients do not have an electronic device or suitable internet connection to receive blended care;
3. Clients have insufficient digital literacy to receive blended care;
4. Families need a translator to receive the intervention.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in Aggression and Delinquency assessed by the Youth Self Report (YSR) | T1 (baseline); monthly during intervention, up to 9 months; T2 (post-intervention) up to 9 months; T3 (follow-up) 6 months post intervention
  The YSR is a self-reported instrument. The Externalizing scale contains 30 items assessing aggression and delinquency. Possible scores range from 0 (never) to 2 (often). For the monthly assessment, a shortened version of the YSR Externalizing scale will be administered.
Change in Aggression and Delinquency assessed with the Child Behavior Checklist (CBCL) | T1 (baseline); monthly during intervention, up to 9 months; T2 (post-intervention) up to 9 months; T3 (follow-up) 6 months post intervention
  The CBCL is a caregiver-reported instrument. The Externalizing scale contains 36 items assessing aggression and delinquency. Possible scores range from 0 (never) to 2 (often). For the monthly assessment, a shortened version of the CBCL Externalizing scale will be administered.
Change in Delinquency assessed with the Self-Report Delinquent Behavior (ZDG) | T1 (baseline); monthly during intervention, up to 9 months; T2 (post-intervention) up to 9 months; T3 (follow-up) 6 months post intervention
  The Self-report Delinquent Behavior [Zelfrapportage Delinquent Gedrag; ZDG] is a self-reported instrument, assessing how many times the juvenile has done certain (rule-breaking) things in the past year. The ZDG contains 30 items. For the monthly assessment, a shortened version of the ZDG will be administered.
Percentage of Participants with Out of Home Placement assessed using File Analysis | T1 (baseline); T2 (post-intervention) up to 9 months
  A participant is viewed as being placed out of home when they do not reside with their primary family, either temporarily or permanently, and either voluntarily or involuntarily. Out of home placement is registered by therapists during treatment as part of the standard FAST procedure.
Percentage of Participants with Out of Home Placement assessed using an Out of Home Placement Questionnaire | T2 (post-intervention) up to 9 months; T3 (follow-up) 6 months post intervention
  A participant is viewed as being placed out of home when they do not reside with their primary family, either temporarily or permanently, and either voluntarily or involuntarily. Out of home placement will be assessed using a questionnaire measuring living situation, which is filled in by juveniles and caregivers. The questionnaire contains one item assessing where the juvenile lives most days of the week.
Change in Recidivism Risk assessed with the RAF GGZ Youth | T1 (baseline); T2 (post-intervention) up to 9 months
  The RAF GGZ Youth is an extensive risk assessment instrument and includes items measuring recidivism risk. The RAF GGZ Youth is filled in by the therapist as part of the standard FAST procedure. Possible scores range from 1 (low) to 5 (high).
Percentage of Participants having Recidivated | T4 (two years post-intervention)
  Recidivism is defined as a conviction, which is coded from official judicial records.

SECONDARY OUTCOMES:
Change in Internalizing Problems assessed with the Youth Self Report (YSR) | T1 (baseline); T2 (post-intervention) up to 9 months; T3 (follow-up) 6 months post intervention
  The YSR is a self-reported instrument. The Internalizing scale contains 31 items, with possible scores ranging from 0 (never) to 2 (often).
Change in Internalizing Problems assessed with the Child Behavior Checklist (CBCL) | T1 (baseline); T2 (post-intervention) up to 9 months; T3 (follow-up) 6 months post intervention
  The CBCL is a caregiver-reported instrument. The Internalizing scale contains 32 items, with possible scores ranging from 0 (never) to 2 (often).
Change in Substance Use assessed with the Monitoring Station Substance Use | T1 (baseline); T2 (post-intervention) up to 9 months; T3 (follow-up) 6 months post intervention
  Monitoring Station Substance Use [Peilstation Middelengebruik] is a self-reported instrument. It contains five items assessing frequency and intensity of substance use.
Change in Substance Use assessed with the RAF GGZ Youth | T1 (baseline); T2 (post-intervention) up to 9 months
  The RAF GGZ Youth is an extensive risk assessment instrument and includes items measuring substance use. The RAF GGZ Youth is filled in by the therapist as part of the standard FAST procedure.
Change in Substance Use assessed with the FAST Goal Lists | T1 (baseline); T2 (post-intervention) up to 9 months
  The FAST Goals Lists are filled in by juveniles, caregivers, and therapists as part of the standard FAST-procedure, and assess the achievement of FAST goals in the past two months. The list includes 1 item on change in substance use. Possible scores range from 1 (not true at all) to 10 (absolutely true).
Change in Contact with Deviant Peers assessed with the Basic Questionnaire Peers (BVL) | T1 (baseline); T2 (post-intervention) up to 9 months; T3 (follow-up) 6 months post intervention
  The Basic Questionnaire Peers [Basisvragenlijst Leeftijdsgenoten; BVL] is a self-reported instrument with 13 items. Possible scores differ per question, for instance measuring amount of friends, or 0 (never) to 4 (5 times or more).
Change in Contact with Deviant Peers assessed with the Family, Friends, & Self Scale (FFSS) | T1 (baseline); T2 (post-intervention) up to 9 months; T3 (follow-up) 6 months post intervention
  The FFSS is a self-reported instrument and contains 16 items. Possible scores range from 1 (none) to 5 (almost all of them).
Change in Client Formulated Goals assessed by the FAST Goal Lists | T1 (baseline); T2 (post-intervention) up to 9 months
  The FAST goal lists are filled in by juveniles, caregivers, and therapists as part of the standard FAST-procedure, and assess the achievement of FAST goals in the past two months. Possible scores range from 1 (not true at all) to 10 (absolutely true).

OTHER OUTCOMES:
Change in Social Support assessed by the Parental Support Questionnaire (PSQ) | T1 (baseline); T2 (post-intervention) up to 9 months; T3 (follow-up) 6 months post intervention
  The PSQ is a caregiver self-reported instrument and contains 15 items. Possible scores range from 0 (no) to 1 (yes), and 1 (unsatisfied) to 5 (satisfied).
Change in Caregiver-Adolescent Conflict assessed by the Network of Relationship Inventory (NRI) | T1 (baseline); monthly from baseline to post intervention, up to 9 months; T2 (post-intervention) up to 9 months; T3 (follow-up) 6 months post intervention
  The NRI is a juvenile and caregiver self-reported instrument. The NRI contains six items with possible scores ranging from 1 (little to not) to 5 (the most). For the monthly assessment, a shortened version of the NRI will be administered.
Change in Caregiver-Adolescent Relationship Quality assessed by the Inventory of Parent and Peer Attachment (IPPA) | T1 (baseline); monthly from baseline to post intervention, up to 9 months; T2 (post-intervention) up to 9 months; T3 (follow-up) 6 months post intervention
  The IPPA is a juvenile self-reported instrument and contains 12 items per caregiver. Possible scores range from 1 (almost never) to 4 (almost always). For the monthly assessment, a shortened version of the IPPA will be administered.
Change in Caregiver-Adolescent Relationship Quality assessed by the Parental Stress Index (NOSI) | T1 (baseline); monthly from baseline to post intervention, up to 9 months; T2 (post-intervention) up to 9 months; T3 (follow-up) 6 months post intervention
  The Parental Stress Index [Nijmeegse Ouderlijke Stress Index; NOSI] is a caregiver self-reported instrument and contains nine items. Possible scores range from 1 (not applicable at all) to 6 (completely applicable). For the monthly assessment, a shortened version of the NOSI will be administered.
Change in Caregiver Responsiveness assessed by the Responsiveness Scale of the Nijmegen Parenting Questionnaire (NOV) | T1 (baseline); monthly from baseline to post intervention, up to 9 months; T2 (post-intervention) up to 9 months; T3 (follow-up) 6 months post intervention
  The Nijmegen Parenting Questionnaire [Nijmeegse Opvoedingsvragenlijst; NOV] is a juvenile and caregiver self-reported instrument. The Responsiveness scale contains eight items. Possible scores range from 1 (completely disagree) to 6 (completely agree). For monthly assessment, a shortened version of the Responsiveness scale will be administered.
Change in Caregiver Consistency assessed by the Consistency Scale of the Nijmegen Parenting Questionnaire (NOV) | T1 (baseline); monthly from baseline to post intervention, up to 9 months; T2 (post-intervention) up to 9 months; T3 (follow-up) 6 months post intervention
  The Nijmegen Parenting Questionnaire [Nijmeegse Opvoedingsvragenlijst; NOV] is a juvenile and caregiver self-reported instrument. The Consistency scale contains eight items. Possible scores range from 1 (completely disagree) to 6 (completely agree). For the monthly assessment, a shortened version of the Consistency scale will be administered.
Change in Behavioral Control assessed by the Parenting Practices | T1 (baseline); monthly from baseline to post intervention, up to 9 months; T2 (post-intervention) up to 9 months; T3 (follow-up) 6 months post intervention
  The Parent Practices is a juvenile and caregiver self-reported instrument and contains six items. Possible scores range from 1 (never) to 5 (always). For the monthly assessment, a shortened version of the Parenting Practices will be administered.
Change in Discipline Practices assessed by the Parenting Dimensions Inventory (PDI) | T1 (baseline); monthly from baseline to post intervention, up to 9 months; T2 (post-intervention) up to 9 months; T3 (follow-up) 6 months post intervention
  The PDI is a juvenile and caregiver self-reported instrument and contains eight items. Possible scores range from 0 (very unlikely) to 3 (very likely). For the monthly assessment, a shortened version of the PDI will be administered.
Change in Psychological Control assessed by the Psychological Control Scale Youth Self-Report (PCS-YSR) | T1 (baseline); monthly from baseline to post intervention, up to 9 months; T2 (post-intervention) up to 9 months; T3 (follow-up) 6 months post intervention
  The PCS-YSR is a self-reported instrument and contains eight items. Possible scores range from 1 (not applicable at all) to 5 (completely applicable). For the monthly assessment, a shortened version of the PCS-YR will be administered.
Change in Caregiver Competence assessed by the Parental Stress Index (NOSI) | T1 (baseline); monthly from baseline to post intervention, up to 9 months; T2 (post-intervention) up to 9 months; T3 (follow-up) 6 months post intervention
  The Parental Stress Index [Nijmeegse Ouderlijke Stress Index; NOSI] is a caregiver self-reported instrument and contains 15 items. Possible scores range from 1 (completely disagree) to 6 (completely agree). For the monthly assessment, a shortened version of the NOSI will be administered.
Change in Cognitive Distortions assessed by the Shortened List Irrational Thoughts (V-LIG) | T1 (baseline); T2 (post-intervention) up to 9 months
  The Shortened List Irrational Thoughts [Verkorte Lijst Irrationele Gedachten; V-LIG] is a self-reported instrument and contains 18 items. Possible scores range from 1 (completely disagree) to 6 (completely agree).
Demographics assessed by a Demographic Information Questionnaire | T1 (baseline)
  The Demographic information questionnaire contains items about gender, age, and occupation. The questionnaire contains nine items for juveniles, 19 for caregivers, and eight for therapists.
Primary Diagnosis assessed by Therapist File Search | T1 (baseline)
  The therapist file contains the primary diagnosis of the juvenile.
Change in Personality assessed by the Inventory of Callous-Unemotional Traits (ICU) | T1 (baseline)
  The ICU is reported by juveniles, caregivers, and therapists and contains 24 items. Possible scores range from 1 (completely untrue) to 4 (always true).
Change in Personality assessed by the Antisocial Process Screening Device (APSD) | T1 (baseline)
  The APSD is reported by juveniles, caregivers, and therapists and contains 12items for juveniles and 16 items for caregivers and therapists. Possible scoresrange from 1 (completely true) to 4 (always true).
Treatment Integrity assessed by the FAST Evaluation Forms | T2 (post-intervention) up to 9 months from baseline
  The FAST evaluation forms are filled in as part of the standard FAST procedure. Possible scores range from 0 (no) to 1 (yes), and 1 (very bad, never) to 10 (very good, always).
Treatment Duration and Intensity assessed by a Treatment Duration and Intensity Questionnaire | T2 (post-intervention) up to 9 months from baseline
  The treatment duration and intensity questionnaire is reported on by the therapist an contains two items. The questionnaire is rated in weeks and average hours per week.
Perceived Treatment Effectiveness assessed by a Perceived Effectiveness Questionnaire | T2 (post-intervention) up to 9 months from baseline
  The perceived effectiveness questionnaire is reported on by the therapist and contains one item. Possible scores range from 1 (sometimes effective) to 4 (almost always effective).
Therapist-Client Alliance assessed by the Relationship with Interventionist | T2 (post-intervention) up to 9 months from baseline
  The Relationship with Interventionist is a juvenile and caregiver self-reported instrument and contains 12 items. Possible scores range from 1 (completely disagree) to 6 (completely agree).
Treatment Satisfaction assessed by the Satisfaction with Program Scale (SPS) | T2 (post-intervention) up to 9 months from baseline
  The SPS is a juvenile and caregiver self-reported instrument and contains 10 items. Possible scores range from 1 (completely disagree) to 6 (completely agree).
Treatment Cooperation assessed by the Cooperation Scale | T2 (post-intervention) up to 9 months from baseline
  The Cooperation Scale is reported on by juveniles, caregivers, and therapists and contains five items. Possible scores range from 1 (completely disagree) to 6 (completely agree).
Treatment Expectancies assessed by the Parent Expectancies for Therapy Scale (PETS) | T1 (baseline)
  The PETS is a caregiver self-reported instrument and contains seven items. Possible scores range from 1 (completely disagree) to 5 (completely agree).
Caregiver Psychopathology assessed by the RAF GGZ Youth | T1 (baseline)
  The RAF GGZ Youth is an extensive risk assessment instrument and includes items measuring caregiver psychopathology. The RAF GGZ Youth is filled in by the therapist as part of the standard FAST procedure. Possible scores range from 0 (problems not present) to 2 (problems definitely present).
Change in Treatment Motivation assessed by the Treatment Motivation Scales for Forensic Outpatient Treatment (TMS-F) | T1 (baseline)
  The TMS-F is reported on by juveniles and caregivers and contains 16 items. Possible scores range from 1 (completely disagree) to 5 (completely agree).

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - de Waag, Utrecht
  - Utrecht University, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
The details on which parts of the data will be shared still have to be discussed.

REFERENCES:
- [Derived] van Cappellen SM, Creemers HE, Hoogsteder L, van Horn J, Dekovic M, Asscher JJ. The effectiveness of blended versus regular Forensic Outpatient Systemic Therapy in the treatment of juvenile antisocial behavior: a study protocol of a randomized controlled trial. BMC Psychiatry. 2023 May 4;23(1):315. doi: 10.1186/s12888-023-04831-8. PMID 37143003
- See also: FAST Intervention Description — https://www.nji.nl/interventies/forensische-ambulante-systeem-therapie-fast